CLINICAL TRIAL: NCT05565248
Title: An Open-Label, First-in-Human Study Evaluating the Safety, Tolerability, and Efficacy of VCTX211 Combination Product in Subjects With Type 1 Diabetes Mellitus (T1D)
Brief Title: An Open-Label, FIH Study Evaluating the Safety, Tolerability, and Efficacy of VCTX211 Combination Product in Subjects With T1D
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CRISPR Therapeutics AG (Industry)
Collaborators: ViaCyte (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCTX211-101
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Type 1 Diabetes; T1D; Allogeneic; Combination Device; CRISPR-Cas9; Cell Therapy; T1DM; Diabetes; VCTX
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VCTX211 unit (Experimental)
  Interventions: Combination Product: VCTX211

INTERVENTIONS:
Combination Product: VCTX211 — CRISPR-Cas9 genetically modified PEC211 cells loaded into a delivery device

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study evaluating the Safety, Tolerability, and Efficacy of VCTX211 Combination Product in Subjects with T1D

DETAILED DESCRIPTION:
VCTX211 combination product (unit) compromises 2 components: (1) allogeneic pancreatic endoderm cells (PEC211) genetically modified using Cluster Regularly Interspaced Short Palindromic Repeats/ CRISPR-associated protein 9 (CRISPR/Cas9) to promote immune evasiveness and survival, and (2) a durable, removable, perforated device designed to deliver and retain PEC211 cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D for a minimum of 5 years
* Stable diabetes regimen for at least 3 months prior to enrollment.

Exclusion Criteria:

* Medical history of islet cell, kidney, and/or pancreas transplant
* Occurrence of 2 or more severe, unexplained hypoglycemic events within 6 months prior to enrollment
* Known causes of diabetes other than T1D
* Immunosuppressant therapy in the previous 30 days and/or requirements for chronic immunosuppressive therapy during the study
* Prior treatment with gene therapy or edited product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events with causality related to VCTX211 units, the surgical procedures and/or medical interventions required to implant and explant the VCTX211 units. | From implantation up to 12 months post implantation
Assess the clinical efficacy of VCTX211 units via evaluation of C-peptide increase from the baseline. | From implantation up to 12 months post implantation

SECONDARY OUTCOMES:
Incidence of adverse events reported in patients implanted with VCTX211 units. | From implantation up to 12 months post implantation
Assess the clinical efficacy of VCTX211 units via evaluation of changes in exogenous insulin use from baseline. | From implantation up to 12 months post implantation
Assess the clinical efficacy of VCTX211 units via evaluation of changes in number of hypoglycemic evens from baseline. | From implantation up to 12 months post implantation
Assess the clinical efficacy of VCTX211 units via evaluation of changes in hemoglobin A1C levels from baseline. | From implantation up to 12 months post implantation
Assess the clinical efficacy of VCTX211 units via evaluation of percentage of time in pre-defined glycemic ranges, as measured by a continuous glucose monitor, from baseline. | From implantation up to 12 months post implantation
Qualitative evaluation of immune response to VCTX211 units assessed by histological staining for markers of host adaptive immune cells within the graft. | From implantation up to 12 months post implantation
Incidence of new alloreactive antibodies found in the blood of patients post implantation. | From implantation up to 12 months post implantation
Incidence of new autoreactive antibodies found in the blood of patients post implantation. | From implantation up to 12 months post implantation
The percentage of viable graft cells per unit using immunohistochemical staining. | From implantation up to 12 months post implantation
The percentage of graft cells per unit that have differentiated into endocrine/beta cells as determined by immunohistochemical staining. | From implantation up to 12 months post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Manasi Jaiman, MD, MPH, Study Director — ViaCyte; Sandeep Soni, MD, Study Director — CRISPR Therapeutics
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia